CLINICAL TRIAL: NCT05646342
Title: PLR in a Good Helath Women After 24 Week of Preganancy
Brief Title: PLR in a Good Helath After 24 Week of Preganancy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Mohammed VI University Hospital (Other)
Responsible Party: Principal Investigator, Younes Oujidi, Doctor, Mohammed VI University Hospital
Other Study IDs: SAR
Record Dates: First submitted 2022-12-05; First posted 2022-12-12 (Actual); Last update posted 2022-12-12 (Actual); Status verified 2022-12

CONDITIONS: ITV Sosu Aortique; Cardiac Output, High; PLR
Keywords: CO; PLR; ETT; Pregnanacy
MeSH Terms: conditions — Cardiac Output, High

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Measure of CO by ECHocardiac Machine — we will realise ETT before and after PLR in all women that eligible of crieria inclusion , in obstetric consultation

SUMMARY:
fluid resuscitation is one of the bases of strategies in ICU to take in charge patients , one of the technique to evaluate preload charge , is Passive leg raising, that allows reliable prediction of fluid responsiveness even in patients with spontaneous breathing activity or arrhythmias .

In recent years, hemodynamic response to passive leg raising (PLR) has been popularized as a dynamic test of preload responsiveness [1]. This manoeuvre provides an "auto-fluid challenge" which is rapid, transient and reversible. PLR transfers blood contained in the venous reservoir of the lower extremities to the central venous compartment leading to a transient increase in preload and an increase in cardiac output by Frank-Starling mechanism in preload responsive individuals.

untille now the usseuful of PLR in Pregnancy, and also The validity of dynamic measurements of preload to predict fluid response during pregnancy are note clear in littérature .

DETAILED DESCRIPTION:
A total of 108 low-risk pregnant women and 54 healthy non-pregnant controls, aged >18 years, participated in the study. Pregnant women attending for the second trimester routine ultrasound screening at 17-19 weeks of gestation were informed about the study and invited to participate if they had a low-risk pregnancy and ultrasound scan did not show any fetal or placental abnormality. Those who agreed were consecutively enrolled and an appointment was made for functional hemodynamic evaluation at 22-24 weeks of gestation. Exclusion criteria were any pre-existing medical condition that may have an effect on the course of pregnancy, and a previous history of preeclampsia, gestational diabetes, intrauterine fetal growth restriction or preterm delivery. Non-pregnant controls were recruited among the nursing, administrative and laboratory staff of the hospital and university. Healthy women of reproductive age were asked to attend for hemodynamic assessment during the follicular phase between day 5 and 10 of the menstrual cycle. Women with a previous history of pregnancy complication and those with a known disease or on regular medication were excluded. Examination was performed,

ELIGIBILITY:
Inclusion Criteria:

* All Pregnante Women in good health after 24 week of preganancy

Exclusion Criteria:

* All young women under 18 years old
* unhealthy women

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Moroccan population
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-04-01 (Estimated)

PRIMARY OUTCOMES:
PLR in a good helath after 24 week of preganancy | in all the 5 mounths
  we will realise ETT before and after PLR in all women that eligible of crieria inclusion , in obstetric consultation

IPD SHARING:
Plan to Share IPD: No